CLINICAL TRIAL: NCT06892834
Title: A Three-month Clinical Study to Assess the Gingivitis Effect of Various Dentifrices.
Brief Title: Assessing Gingivitis of 3 Different Dentifrices Compared to a Negative Control.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024026
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Positive Control (Active Comparator): 0.454% stannous fluoride, 0.533% zinc citrate
  Interventions: Drug: Stannous Fluoride Dentifrice
- Experimental #1 (Experimental): 0.243% NaF with 0.1% Hops, Humulus lupulus extract [0.045% hops β-acids]
  Interventions: Drug: Sodium Fluoride Dentifrice
- Experimental #2 (Experimental): 0.243% NaF with 0.5% Hops, Humulus lupulus extract [0.225% hops β-acids]
  Interventions: Drug: Sodium Fluoride Dentifrice
- Negative Control (Active Comparator): 0.76% Sodium Monofluorophosphate
  Interventions: Drug: Sodium monofluorophosphate dentifrice

INTERVENTIONS:
Drug: Stannous Fluoride Dentifrice — Each subject will be randomly assigned to one of four treatment products and will be asked to brush 2x a day (1 minute per brushing) for 3 months.
  Arms: Positive Control
Drug: Sodium Fluoride Dentifrice — Each subject will be randomly assigned to one of four treatment products and will be asked to brush 2x a day (1 minute per brushing) for 3 months.
  Arms: Experimental #1; Experimental #2
Drug: Sodium monofluorophosphate dentifrice — Each subject will be randomly assigned to one of four treatment products and will be asked to brush 2x a day (1 minute per brushing) for 3 months.
  Arms: Negative Control

SUMMARY:
The primary objective of this study is to evaluate the effect of two experimental hops extract-containing dentifrices on gingivitis relative to a positive control 0.454% SnF2 dentifrice and a negative control dentifrice after 12 weeks of product use.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial; If female of child-bearing potential, agree to use a medically approved method of birth control for the duration of the study. Acceptable methods of medically approved birth control include: at least 3 months of use of a hormonal birth control (including oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant), double-barrier method, intrauterine devices, non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s), vasectomy of partner at least 6 months prior to screening. Not applicable to females not of child-bearing potential (females who have undergone a sterilization procedure including hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior;
* If female and of child-bearing potential, agree to immediately inform the study investigator if they become pregnant;
* Have at least 20 gradable teeth;
* Have mild to moderate gingivitis with a range of 10 to 70% bleeding sites;
* Agree to return for scheduled visits and follow the study procedures;
* Agree to refrain from use of any non-study oral hygiene products for the duration of the study; regular floss users can continue to floss in their customary manner.
* Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study; and
* Agree to refrain from any oral hygiene the morning of each visit.

Exclusion Criteria:

* Having taken antibiotic, anti-inflammatory, or anticoagulant medications within 4 weeks of the baseline visit;
* Having any oral conditions that could interfere with study compliance and/or examination procedures, such as widespread caries, soft or hard tissue tumor of the oral cavity, severe gingivitis, or advanced periodontal disease;
* Females of child-bearing potential who are not using a medically approved method of birth control (i.e., hormonal contraceptives including oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant, double-barrier method, intrauterine devices, non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s), vasectomy of partner at least 6 months prior to screening) or who have not been using hormonal birth control for a minimum of 3 months prior to study enrollment;
* Taking medication that alters gingival appearance or gingival bleeding (e.g., calcium channel blockers, anticonvulsants, or immunosuppressants) within one month prior to study initiation;
* Regularly (>5x/week) using anti-gingivitis treatments (e.g., stannous fluoride toothpaste, or anti-gingivitis mouthwashes, such as those containing chlorohexidine) in the month prior to screening;
* Removable oral appliances;
* Fixed facial or lingual orthodontic appliances;
* Have a positive pregnancy test (Clearblue) at baseline or self-reported pregnancy during the study; ;
* Any diseases or condition that might interfere with the safe participation in the study according to the study investigator;
* Inability to undergo study procedures; and
* Allergic reactions to any of the study toothpastes and/or ingredients in the study toothpastes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Number Bleeding Sites | 1 month and 3 months

SECONDARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | 1 month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: All Sum Research, Principal Investigator — All Sum Research
Locations (1):
- All Sum ResearchAll Sum Research Center Ltd., Mississauga, Ontario, Canada